CLINICAL TRIAL: NCT02141438
Title: Radium-223 Alpha Emitter Agent in Non-intervention Safety Study in mCRPC popUlation for Long-teRm Evaluation
Brief Title: Observational Study for the Evaluation of Long-term Safety of Radium-223 Used for the Treatment of Metastatic Castration Resistant Prostate Cancer
Acronym: REASSURE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16913
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Results first posted 2025-09-05 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Radium-223; CRPC; Phase IV; Safety study
MeSH Terms: interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radium-223 dichloride (Xofigo, BAY88-8223): Single-arm cohort observational study with CRPC patients with bone metastasis treated with Radium-223.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — This is a non-interventional study, the drug is used in its authorized indication from commercial supply. The decision to treat with Radium-223 will be agreed upon between the physician and the patient independently and prior to providing the patient study information. Treatment with Radium-223 should follow the approved local product information.

SUMMARY:
Observational study in the routine clinical practice setting to evaluate the short and long term safety profile of Radium-223 in metastatic castration resistant prostate cancer patients and to evaluate the risk of developing second primary cancers.

ELIGIBILITY:
Inclusion Criteria:

* Treatment decision to Radium-223 needs to be made independent from and before patient enrollment in the study
* Histologically or cytologically confirmed castration resistant adenocarcinoma of the prostate with bone metastases
* Signed informed consent

Exclusion Criteria:

* Previously treated with Radium-223 for any reason
* Currently treated in clinical trials including other Radium-223 studies
* Planned for the systemic concomitant use of other radiopharmaceuticals for treatment of prostate cancer or for other use

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed castration resistant adenocarcinoma of the prostate with bone metastases for whom the treatment decision to Radium-223 has been made independent from and before patient enrolment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1472 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (68):
- United States (49):
  - Anchorage, Alaska
  - Scottsdale, Arizona
  - Daly City, California
  - Long Beach, California
  - Sacramento, California
  - San Diego, California
  - Colorado Springs, Colorado
  - Boca Raton, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Lakewood Rch, Florida
  - Plantation, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Honolulu, Hawaii
  - Evanston, Illinois
  - Warrenville, Illinois
  - Wichita, Kansas
  - Ashland, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Rockville, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Troy, Michigan
  - St Louis, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Neptune City, New Jersey
  - Township, New Jersey
  - Buffalo, New York
  - East Setauket, New York
  - Lake Success, New York
  - Winston-Salem, North Carolina
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Springfield, Oregon
  - Abington, Pennsylvania
  - Charleston, South Carolina
  - Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - Lubbock, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Charlottesville, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington
- Multiple Locations, Argentina
- Multiple Locations, Austria
- Multiple Locations, Belgium
- Multiple Locations, Canada
- Multiple Locations, Colombia
- Multiple Locations, Czechia
- Multiple Locations, Denmark
- Multiple Locations, France
- Multiple Locations, Germany
- Multiple Locations, Greece
- Multiple Locations, Israel
- Multiple Locations, Italy
- Multiple Locations, Luxembourg
- Multiple Locations, Mexico
- Multiple Locations, Netherlands
- Multiple Locations, Portugal
- Multiple Locations, Spain
- Multiple Locations, Sweden
- Multiple Locations, United Kingdom

REFERENCES:
- [Derived] O'Sullivan JM, Heinrich D, Castro E, George S, Dizdarevic S, Baldari S, Essler M, Jong IJ, Lastoria S, Hammerer PG, Tombal B, James ND, Meltzer J, Sandstrom P, Sartor O. Alkaline phosphatase decline and pain response as predictors of overall survival benefit in patients treated with radium-223: a post hoc analysis of the REASSURE study. Br J Cancer. 2025 Mar;132(4):354-360. doi: 10.1038/s41416-024-02927-w. Epub 2025 Jan 9. PMID 39789153
- [Derived] Higano CS, Dizdarevic S, Logue J, Richardson T, George S, de Jong I, Tomaszewski JJ, Saad F, Miller K, Meltzer J, Sandstrom P, Verholen F, Tombal B, Sartor O. Safety and effectiveness of the radium-223-taxane treatment sequence in patients with metastatic castration-resistant prostate cancer in a global observational study (REASSURE). Cancer. 2024 Jun 1;130(11):1930-1939. doi: 10.1002/cncr.35221. Epub 2024 Feb 10. PMID 38340349
- [Derived] Sartor O, Fougere C, Essler M, Ezziddin S, Kramer G, Ellinger J, Nordquist L, Sylvester J, Paganelli G, Peer A, Bogemann M, Meltzer J, Sandstrom P, Verholen F, Song DY. 177Lu-Prostate-Specific Membrane Antigen Ligand After 223Ra Treatment in Men with Bone-Metastatic Castration-Resistant Prostate Cancer: Real-World Clinical Experience. J Nucl Med. 2022 Mar;63(3):410-414. doi: 10.2967/jnumed.121.262240. Epub 2021 Jun 24. PMID 34168015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 188 treatment centers in 20 countries from 20 August 2014 (first patient first visit) to 02 August 2024 (last patient last visit)
Pre-assignment Details: Overall, 1567 participants were screened and a total of 1472 participants started treatment with Radium-223
Groups:
- Radium-223: Participants with castration-resistant prostate cancer (CRPC) with bone metastases have received Radium-223 as part of their routine care at participating study centers
Period: Overall Study
Arm/Group | Radium-223
Started | 1472
Completed | 22
Not Completed | 1450
Not completed — Death | 1308
Not completed — Lost to Follow-up | 84
Not completed — Withdrawal by Subject | 52
Not completed — Physician Decision | 1
Not completed — Patients without documented end of observation due to premature site closure | 5

BASELINE CHARACTERISTICS:
Arm/Group | Radium-223
Number analyzed (Participants) | 1472
Age, Continuous [Median (Full Range); unit: Years] | 73.0 [44 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1472
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 170
  Not Hispanic or Latino | 1159
  Unknown or Not Reported | 143
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1295
  Black or African American | 63
  Asian | 16
  Multiple | 2
  American Indian or Alaska Native | 1
  Not reported | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Second Primary Malignancies (SPM)
Description: Second primary malignancies (SPMs) are defined as new malignancies unrelated to prostate cancer or progression of prostate cancer. All types of SPMs will be collected irrespectively of their relationship to Radium-223. All reported SPMs will be summarized as assessed by the physician
Time Frame: From the initiation of Radium-223 (treatment period up to 6 months which includes 6 cycles every 4 weeks) up to 7 years after the last dose of Radium-223
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223
Number analyzed (Participants) | 1472
Participants | 24

2. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: Treatment-emergent was defined as any event arising or worsening on the day of or after start of radium-223 until 30 days after last injection.
Time Frame: From initiation of Radium-223 (treatment period up to 6 months which includes 6 cycles every 4 weeks) up to 30 days after the last administration of Radium-223
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223
Number analyzed (Participants) | 1472
Participants | 325

3. Primary Outcome: Number of Participants With Drug-related Treatment-emergent Adverse Events
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223
Number analyzed (Participants) | 1472
Participants | 537

4. Primary Outcome: Number of Participants With Drug-related SAEs
Description: All drug-related SAEs were collected up to 7 years after the last administration of radium-223.
Time Frame: From initiation of Radium-223 (treatment period up to 6 months which includes 6 cycles every 4 weeks), up to 7 years after the last dose of Radium-223
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223
Number analyzed (Participants) | 1472
Participants | 88

5. Primary Outcome: Number of Participants With Therapeutic or Preventive Treatments for Bone Marrow Suppression
Description: Bone marrow suppression relevant treatments for participants with subsequent chemotherapy (e.g., blood transfusion/erythropoietin/colony growth stimulating factors)
Time Frame: From initiation of Radium-223 (treatment period up to 6 months which includes 6 cycles every 4 weeks) up to 6 months after last dose of Radium-223
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223
Number analyzed (Participants) | 1472
Participants
  Patients with at least one of the bone marrow suppression relevant treatments: No | 1133
  Patients with at least one of the bone marrow suppression relevant treatments: Yes | 339
  Patients with any blood transfusions: No | 1155
  Patients with any blood transfusions: Yes | 317
  Patients receiving erythropoiesis stimulating drugs: No | 1448
  Patients receiving erythropoiesis stimulating drugs: Yes | 24
  Patients with colony stimulating factors: No | 1448
  Patients with colony stimulating factors: Yes | 24

6. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time interval from the start of Radium-223 therapy to death due to any cause. Patients whose death was not confirmed at the time of data-cut were censored at the last date known to be alive.
Time Frame: From initiation of Radium-223 (treatment period up to 6 months which includes 6 cycles every 4 weeks) up to 7 years after the last dose of Radium-223
Population: Safety analysis set (SAF)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223
Number analyzed (Participants) | 1472
Months | 15.6 [14.6 to 16.4]

7. Secondary Outcome: Worst Pain Score Over Time as Determined by Patient Responses on the "Brief Pain Inventory Short Form" (BPI-SF) Questionnaire
Description: The Brief pain inventory short form (BPI-SF) questionnaire was used to assess pain severity on a scale from 0 (no pain) to 10 (worst pain). The BPI-SF questionnaire was requested prior to each injection of Radium-223 and also used at each follow-up visit until 6 months after the last injection of Radium-223. The pain severity score was calculated per visit. Completion of the BPI-SF questionnaire by the patient was voluntary. Since this is an observational study, the treatment regimen may not necessarily follow the recommended schedule of one cycle every 4 weeks for all participants
Time Frame: From initiation of Radium-223 (treatment period up to 6 months which includes 6 cycles every 4 weeks) up to 6 months after the last dose of Radium-223
Population: Safety analysis set (SAF)
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Radium-223
Number analyzed (Participants) | 1356
Score
  Baseline/Treatment cycle 1 | 3.003 (2.189)
  Treatment cycle 2 (approximately at week 4): number analyzed (Participants) | 1182
  Treatment cycle 2 (approximately at week 4) | 2.760 (2.251)
  Treatment cycle 3 (approximately at week 8): number analyzed (Participants) | 1090
  Treatment cycle 3 (approximately at week 8) | 2.464 (2.222)
  Treatment cycle 4 (approximately at week 12): number analyzed (Participants) | 943
  Treatment cycle 4 (approximately at week 12) | 2.436 (2.309)
  Treatment cycle 5 (approximately at week 16): number analyzed (Participants) | 828
  Treatment cycle 5 (approximately at week 16) | 2.261 (2.223)
  Treatment cycle 6 (approximately at week 20): number analyzed (Participants) | 736
  Treatment cycle 6 (approximately at week 20) | 2.262 (2.210)
  First available follow-up measurement: number analyzed (Participants) | 502
  First available follow-up measurement | 2.458 (2.307)
  Last available follow-up measurement: number analyzed (Participants) | 502
  Last available follow-up measurement | 2.629 (2.424)

8. Secondary Outcome: The Pain Interference Score Over Time as Determined by Patient Responses on the "Brief Pain Inventory Short Form" (BPI-SF) Questionnaire
Description: The Brief pain inventory short form (BPI-SF) questionnaire was used to assess pain interference on a scale from 0 (does not interfere) to 10 (completely interferes). The BPI-SF questionnaire was requested prior to each injection of Radium-223 and also used at each follow-up visit until 6 months after the last injection of Radium-223. The pain interference score was calculated per visit. Completion of the BPI-SF questionnaire by the patient was voluntary Since this is an observational study, the treatment regimen may not necessarily follow the recommended schedule of one cycle every 4 weeks for all participants
Time Frame: From initiation of Radium-223 (treatment period up to 6 months which includes 4 cycles every 4 weeks) up to 6 months after the last dose of Radium-223
Population: Safety analysis set (SAF)
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Radium-223
Number analyzed (Participants) | 1364
Score
  Baseline/Treatment 1 | 3.283 (2.664)
  Treatment cycle 2 (approximately at week 4): number analyzed (Participants) | 1185
  Treatment cycle 2 (approximately at week 4) | 2.965 (2.588)
  Treatment cycle 3 (approximately at week 8): number analyzed (Participants) | 1091
  Treatment cycle 3 (approximately at week 8) | 2.656 (2.469)
  Treatment cycle 4 (approximately at week 12): number analyzed (Participants) | 937
  Treatment cycle 4 (approximately at week 12) | 2.587 (2.525)
  Treatment cycle 5 (approximately at week 16): number analyzed (Participants) | 826
  Treatment cycle 5 (approximately at week 16) | 2.358 (2.408)
  Treatment cycle 6 (approximately at week 20): number analyzed (Participants) | 736
  Treatment cycle 6 (approximately at week 20) | 2.495 (2.425)
  First available follow-up measurement: number analyzed (Participants) | 503
  First available follow-up measurement | 2.809 (2.570)
  Last available follow-up measurement: number analyzed (Participants) | 504
  Last available follow-up measurement | 3.107 (2.774)

9. Secondary Outcome: Percentage of Participants With Bone Fractures
Description: Bone fractures were identified by MedDRA HLGTs: Fractures: HLGT = "Fractures".
Time Frame: From initiation of Radium-223 (treatment period up to 6 months which includes 6 cyles every 4 weeks) up to 7 years post last dose of Radium-223
Population: Safety analysis set (SAF)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Radium-223
Number analyzed (Participants) | 1472
Percentage of participants | 9.7 [8.2 to 11.3]

10. Secondary Outcome: Percentage of Participants With Bone Associated Events
Description: Bone associated events were identified by MedDRA HLGTs: Bone associated events: HLGT = "Bone disorders (excl congenital and fractures)"
Time Frame: as for outcome 9
Population: Safety analysis set (SAF)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Radium-223
Number analyzed (Participants) | 1472
Percentage of participants | 8.5 [7.1 to 10.0]

11. Primary Outcome: Incidences of Post-Radium-223 Treatment CTCAE Grade 3/4 Hematological Toxicities Based on Bone Marrow Suppression
Description: Hematological toxicities were summarized by the Common Terminology Criteria for Adverse Events (CTCAE) coding system and the worst grade. The grading system ranges from Grade 1 (mild) to Grade 5 (death). The percentage of participants with post-radium-223 treatment CTCAE grade 3 or 4 hematological toxicities that occurred within 183 days from last radium-223 injection are reported
Time Frame: From last Radium-223 dose up to 6 months post last dose of Radium-223
Population: Safety analysis set (SAF)
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Radium-223
Number analyzed (Participants) | 1472
Percentage
  Grade 3 | 14.74 [12.97 to 16.66]
  Grade 4 | 1.77 [1.16 to 2.58]
  Total | 15.42 [13.61 to 17.37]

12. Primary Outcome: Bone Marrow Suppression: Number of Participants With Abnormal Platelet Count or White Blood Cell Count (WBC)
Description: Participants with a platelet count or WBC less than the lower limit of normal at 6 months post last dose of Radium- 223
Time Frame: From 30 days after last dose of Radium-223 up to 6 months after last dose
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223
Number analyzed (Participants) | 1472
Participants
  Abnormal platelet count (<50x10^9/L): No | 398
  Abnormal platelet count (<50x10^9/L): Yes | 49
  Abnormal platelet count (<50x10^9/L): Missing | 1025
  Abnormal neutrophil count (<1x10^9/L): No | 247
  Abnormal neutrophil count (<1x10^9/L): Yes | 6
  Abnormal neutrophil count (<1x10^9/L): Missing | 1219

13. Primary Outcome: Bone Marrow Suppression: Number of Participants Who Underwent Subsequent Chemotherapy That Experienced Febrile Neutropenia or Hemorrhage
Description: Participants who receive subsequent cytotoxic chemotherapy were followed for the development of febrile neutropenia and hemorrhage up to 6 months after the last administration of chemotherapy at a frequency based on local clinical practice.
Time Frame: From first dose of subsequent chemotherapy up to 6 months (up to 183 days) after the last administration of chemotherapy
Population: Safety analysis set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223
Number analyzed (Participants) | 391
Participants | 23

ADVERSE EVENTS:
Time Frame: After initiation of Radium-223 (treatment period up to 6 months which includes 6 cycles every 4 weeks) up to 30 days after the last administration of Radium-223. Drug-related serious adverse events were collected up to 7 years. Adverse events reporting for all-cause mortality considers all death that occurred at any time during the study before the last contact, up to 7 years after last administration of Radium-223.
Description: Drug-related treatment-emergent adverse events (TEAEs)
Arm/Group | Radium-223
All-Cause Mortality (participants affected / at risk) | 1308/1472
Serious Adverse Events (participants affected / at risk) | 325/1472
Other Adverse Events (participants affected / at risk) | 837/1472
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 (N=1472)
Anaemia (Blood and lymphatic system disorders) | 27 (30)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3)
Angina pectoris (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (6)
Cardiac failure (Cardiac disorders) | 6 (6)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2)
Cardiovascular disorder (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (1)
Papilloedema (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 8 (8)
Chest pain (General disorders) | 3 (3)
Condition aggravated (General disorders) | 1 (1)
Death (General disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Hyperthermia (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 10 (11)
Pyrexia (General disorders) | 5 (5)
Swelling face (General disorders) | 1 (1)
Performance status decreased (General disorders) | 3 (3)
Peripheral swelling (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 15 (15)
Inflammation (General disorders) | 1 (1)
Disease progression (General disorders) | 4 (4)
Multiple organ dysfunction syndrome (General disorders) | 4 (4)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 4 (4)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (3)
Mastoiditis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 14 (14)
Pyelonephritis (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 5 (5)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (7)
Viral infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 5 (5)
Groin abscess (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (3)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 5 (5)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 4 (4)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1)
Full blood count decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 5 (7)
International normalised ratio increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 6 (6)
Red blood cell count decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 2 (2)
Cachexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukaemia monocytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (16)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Hormone-refractory prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 4 (4)
Cerebrovascular accident (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Monoparesis (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 13 (14)
Superior sagittal sinus thrombosis (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Balance disorder (Nervous system disorders) | 1 (1)
IIIrd nerve paresis (Nervous system disorders) | 1 (1)
Intracranial haematoma (Nervous system disorders) | 1 (1)
Spinal cord disorder (Nervous system disorders) | 1 (1)
Epidural lipomatosis (Nervous system disorders) | 1 (1)
Intracranial mass (Nervous system disorders) | 1 (2)
Medullary compression syndrome (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 5 (5)
Hydronephrosis (Renal and urinary disorders) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3)
Ureteric stenosis (Renal and urinary disorders) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 6 (6)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (6)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Disability (Social circumstances) | 1 (1)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1)
Shoulder operation (Surgical and medical procedures) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Pelvic venous thrombosis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 (N=1472)
Anaemia (Blood and lymphatic system disorders) | 168 (193)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 20 (21)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 21 (22)
Pancytopenia (Blood and lymphatic system disorders) | 6 (6)
Pernicious anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 37 (37)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1)
Haematotoxicity (Blood and lymphatic system disorders) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Cardiac failure (Cardiac disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 5 (6)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Exophthalmos (Eye disorders) | 1 (1)
Retinal tear (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 11 (11)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 12 (14)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Change of bowel habit (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 49 (51)
Diarrhoea (Gastrointestinal disorders) | 203 (270)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 10 (10)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Eructation (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 4 (4)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 2 (2)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 189 (212)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 67 (79)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 1 (1)
Mouth swelling (Gastrointestinal disorders) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 4 (4)
Asthenia (General disorders) | 62 (68)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 10 (10)
Chills (General disorders) | 4 (4)
Discomfort (General disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 170 (182)
Feeling cold (General disorders) | 1 (1)
Gait disturbance (General disorders) | 3 (3)
Influenza like illness (General disorders) | 6 (6)
Injection site haemorrhage (General disorders) | 1 (1)
Malaise (General disorders) | 5 (5)
Mass (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 3 (3)
Oedema (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 30 (31)
Pain (General disorders) | 55 (56)
Pyrexia (General disorders) | 16 (22)
Performance status decreased (General disorders) | 2 (2)
Peripheral swelling (General disorders) | 7 (7)
General physical health deterioration (General disorders) | 9 (9)
Temperature intolerance (General disorders) | 1 (1)
Early satiety (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Illness (General disorders) | 2 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (2)
Abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3)
Conjunctivitis (Infections and infestations) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (2)
Ear infection (Infections and infestations) | 2 (2)
Erysipelas (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (3)
Herpes zoster (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 4 (4)
Labyrinthitis (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 5 (6)
Nasopharyngitis (Infections and infestations) | 8 (8)
Onychomycosis (Infections and infestations) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (3)
Otitis externa (Infections and infestations) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Skin infection (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urethritis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 14 (14)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Spinal cord infection (Infections and infestations) | 3 (3)
Escherichia urinary tract infection (Infections and infestations) | 2 (2)
Helicobacter gastritis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Herpes dermatitis (Infections and infestations) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 15 (18)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2)
Ilium fracture (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 5 (5)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 3 (3)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (4)
Chest injury (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood calcium decreased (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 5 (6)
Blood glucose increased (Investigations) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 26 (40)
International normalised ratio increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 11 (15)
Neutrophil count decreased (Investigations) | 12 (13)
Platelet adhesiveness increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 20 (21)
Prostatic specific antigen increased (Investigations) | 4 (4)
Protein total decreased (Investigations) | 1 (2)
Red blood cell count decreased (Investigations) | 2 (2)
Weight decreased (Investigations) | 36 (46)
Weight increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 22 (26)
Blood glucose fluctuation (Investigations) | 1 (2)
Ejection fraction decreased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 8 (8)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 (1)
Intestinal transit time decreased (Investigations) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 13 (13)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2)
Food aversion (Metabolism and nutrition disorders) | 1 (1)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 85 (86)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 73 (89)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 86 (95)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 55 (56)
Coccydynia (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 5 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 12 (12)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Myopathy (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 43 (49)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Sacral pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 14 (15)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 5 (5)
Spinal pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Jaw fistula (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Amnesia (Nervous system disorders) | 2 (2)
Areflexia (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 17 (18)
Dysgeusia (Nervous system disorders) | 12 (12)
Headache (Nervous system disorders) | 20 (21)
Hypersomnia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 4 (4)
Hypogeusia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 10 (10)
Memory impairment (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 19 (20)
Parosmia (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 9 (9)
Somnolence (Nervous system disorders) | 6 (6)
Spinal cord compression (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 5 (5)
Tremor (Nervous system disorders) | 3 (3)
Trigeminal neuralgia (Nervous system disorders) | 2 (2)
Balance disorder (Nervous system disorders) | 2 (2)
Intercostal neuralgia (Nervous system disorders) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Neurological decompensation (Nervous system disorders) | 1 (1)
Taste disorder (Nervous system disorders) | 5 (5)
Brain fog (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Bruxism (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 5 (5)
Depressed mood (Psychiatric disorders) | 5 (5)
Depression (Psychiatric disorders) | 5 (5)
Hallucination (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (6)
Restlessness (Psychiatric disorders) | 1 (1)
Calculus urethral (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 4 (4)
Haematuria (Renal and urinary disorders) | 17 (20)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Nocturia (Renal and urinary disorders) | 4 (4)
Pollakiuria (Renal and urinary disorders) | 7 (7)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Urethral obstruction (Renal and urinary disorders) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 5 (5)
Urinary retention (Renal and urinary disorders) | 3 (3)
Urinary tract disorder (Renal and urinary disorders) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 1 (1)
Bladder mass (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 6 (8)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 3 (3)
Genital erythema (Reproductive system and breast disorders) | 1 (1)
Pelvic discomfort (Reproductive system and breast disorders) | 1 (1)
Penile oedema (Reproductive system and breast disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (24)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Madarosis (Skin and subcutaneous tissue disorders) | 1 (1)
Bedridden (Social circumstances) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 9 (9)
Lymphoedema (Vascular disorders) | 3 (3)
Poor peripheral circulation (Vascular disorders) | 1 (1)
Systolic hypertension (Vascular disorders) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Hot flush (Vascular disorders) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall not publish results of the study before the first multi-center publication, unless agreed otherwise. If no multi-center publication occurs within 18 months after study completion, the PI may publish results at their site, provided they submit the publication to the sponsor at least 60 days prior for review and delay publication for up to 60 days if advised by the sponsor regarding patentable subject matter or Confidential Information (CI) to allow for patent filing or CI removal

DOCUMENTS (2):
  • Study Protocol (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT02141438/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT02141438/SAP_001.pdf